CLINICAL TRIAL: NCT06710314
Title: A Metabolomics-based Study to Explore the Mechanism of Remission of Metabolic Syndrome Radical Resection of Colorectal Cancer
Status: Enrolling by invitation | Type: Observational
Sponsor: Dong Peng (Other)
Responsible Party: Sponsor-Investigator, Dong Peng, First Affiliated Hospital of Chongqing medical university, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Other Study IDs: Chongqing Medical University
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Metabolomics
Keywords: colorectal cancer; Metabolomics; hypertension; diabetes; fatty liver
MeSH Terms: conditions — Colorectal Neoplasms; Hypertension; Diabetes Mellitus; Fatty Liver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Diagnostic Test：Hypertension: Hypertension
  Interventions: Diagnostic Test: Colorectal cancer patients with hypertension
- Diagnostic Test：Diabetes: Diabetes
  Interventions: Diagnostic Test: Colorectal cancer patients with diabetes
- Diagnostic Test：fatty liver: fatty liver
  Interventions: Diagnostic Test: Colorectal cancer patients with fatty liver

INTERVENTIONS:
Diagnostic Test: Colorectal cancer patients with hypertension — Colorectal cancer patients with hypertension
  Groups: Diagnostic Test：Hypertension
Diagnostic Test: Colorectal cancer patients with diabetes — Colorectal cancer patients with diabetes
  Groups: Diagnostic Test：Diabetes
Diagnostic Test: Colorectal cancer patients with fatty liver — Colorectal cancer patients with fatty liver
  Groups: Diagnostic Test：fatty liver

SUMMARY:
1. Analysis of preoperative and postoperative metabolite changes: Through metabolomics technology, the changes of preoperative and postoperative metabolites in patients with colorectal cancer complicated with metabolic syndrome such as hypertension and diabetes were systematically analyzed, and the key metabolites related to postoperative remission were found.
2. Explore the influencing factors of postoperative remission of metabolic syndrome: Combined with clinical data, the association between various metabolites and the degree of postoperative remission was evaluated, and the main factors affecting postoperative remission were determined.

To reveal the mechanism of the remission of metabolic syndrome after surgery: To clarify the metabolic pathways and mechanisms involved in the remission of metabolic syndrome after surgery through multi-level metabolomics analysis, and to provide a new theoretical basis for the development of tumor metabolic surgery.

DETAILED DESCRIPTION:
This study will continue for 2-3 years. All patients who meet the inclusion and exclusion criteria will be divided into hypertension group and diabetes group according to the type of metabolic syndrome, with 120 cases in each group. Blood and feces of all patients were collected before surgery, 3 days after surgery, 6 months after surgery, and 1 year after surgery. The collected samples will be subjected to untargeted metabolomics analysis, using NMR-IVDr technology to detect the dynamic changes of all small molecular metabolites (mainly endogenous small molecular compounds with relative molecular weight within 1000 Da) in blood and feces before and after stimulation or disturbance without bias. The differential metabolites of blood glucose, blood lipids, cholesterol, insulin, renin, aldosterone and angiotensin were screened by bioinformatics analysis, and the pathway analysis of differential metabolites was performed to reveal the potential physiological mechanism of postoperative hypertension, diabetes and other metabolic syndrome remission

ELIGIBILITY:
Inclusion Criteria:

* 1. Age >18 years old. 2. Patients with hypertension or diabetes for more than 1 year before surgery. 3. Patients who planned to undergo radical resection of colorectal cancer

Exclusion Criteria:

* 1. Emergency operation due to intestinal obstruction and intestinal perforation. 2. Tumor with distant metastasis. 3. Combined resection of other important organs. 4. Severe postoperative complications. 5. Patients who are using drugs that may significantly affect metabolic status (such as hormonal drugs, potent immunosuppressants, etc.). 6. Incomplete clinical data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Colorectal cancer complicated with metabolic syndrome such as hypertension, diabetes and fatty liver
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Metabolic disease remission | From date of surgery until the date of first documented postoperative complication, assessed up to 2 months after surgery.
  Metabolic disease remission was defined as any remission of hypertention, diabetes, or fatty liver measured 2 months after surgery. Hypertension remission was defined as arterial blood pressure less than 140/90 mmHg measured postoperatively in patients with preoperative comorbid hypertension. Diabetes remission was defined as fasting blood glucose less than 6 mmol/L measured postoperatively in patients with preoperative comorbid diabetes. Fatty liver remission was defined as liver function in the normal range measured by postoperative blood tests in patients with preoperative comorbid fatty liver.

CONTACTS AND LOCATIONS:
Locations (1):
- Chongqing medical university, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing was not permitted at the performing clinical sites

REFERENCES:
- [Background] Peng D, Liu XY, Cheng YX, Tao W, Cheng Y. Improvement of Diabetes Mellitus After Colorectal Cancer Surgery: A Retrospective Study of Predictive Factors For Type 2 Diabetes Mellitus Remission and Overall Survival. Front Oncol. 2021 Jul 6;11:694997. doi: 10.3389/fonc.2021.694997. eCollection 2021. PMID 34295822
- [Background] Cheng HC, Chang TK, Su WC, Tsai HL, Wang JY. Narrative review of the influence of diabetes mellitus and hyperglycemia on colorectal cancer risk and oncological outcomes. Transl Oncol. 2021 Jul;14(7):101089. doi: 10.1016/j.tranon.2021.101089. Epub 2021 Apr 7. PMID 33838541
- [Background] Petrelli F, Ghidini M, Rausa E, Ghidini A, Cabiddu M, Borgonovo K, Ghilardi M, Parati MC, Pietrantonio F, Sganzerla P, Bossi AC. Survival of Colorectal Cancer Patients With Diabetes Mellitus: A Meta-Analysis. Can J Diabetes. 2021 Mar;45(2):186-197.e2. doi: 10.1016/j.jcjd.2020.06.009. Epub 2020 Jun 20. PMID 33039329
- [Background] Ricci C, Gaeta M, Rausa E, Macchitella Y, Bonavina L. Early impact of bariatric surgery on type II diabetes, hypertension, and hyperlipidemia: a systematic review, meta-analysis and meta-regression on 6,587 patients. Obes Surg. 2014 Apr;24(4):522-8. doi: 10.1007/s11695-013-1121-x. PMID 24214202
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593